CLINICAL TRIAL: NCT02423538
Title: A Phase I, Randomized, Placebo-Controlled, Single Dose Escalation Study to Investigate Safety, Pharmacokinetics and Pharmacodynamics of SHR0302 in Healthy Volunteers
Brief Title: First-in-Human Single Ascending Dose of SHR0302
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR0302-101
Record Dates: First submitted 2015-04-07; First posted 2015-04-22 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ivarmacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- single ascending doses (Experimental): single ascending doses, oral tablets
  Interventions: Drug: SHR0302
- Placebo (Placebo Comparator): Placebo Comparator, oral tablets
  Interventions: Drug: SHR0302 placebo comparator

INTERVENTIONS:
Drug: SHR0302 — Oral tablets (1 mg, 5 mg, 10 mg)
  Arms: single ascending doses
Drug: SHR0302 placebo comparator — Oral tablets (1 mg, 5 mg, 10 mg) (matching corresponding study medication)
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of single ascending (SAD) oral doses of SHR0302 compared to placebo. Also, pharmacokinetics (PK) and pharmacodynamics (PD) of SHR0302 after single oral administration will be evaluated, and, if applicable, the maximum tolerated dose determined.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, age 18-45 years (inclusive);
* The weight of the subject should be more than 50 kg, body mass index (BMI = weight/height squared (kg/m2)) within the range of 19 to 24.

Exclusion Criteria:

* Any condition that might interfere with the procedures or tests in the study
* History of heart failure or renal insufficiency
* Smoking; Drug or alcohol abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Adverse events and the number of volunteers with adverse events as a measure of safety and tolerability. | up to 72 hrs postdose
  Tests will be performed to assess whether the study drug has any potentially adverse effect (laboratory tests on blood and urine for functioning of organs; cardiovascular testing, i.e. of heart and blood circulation). Also, participants will carefully be monitored by medical staff for vital signs, and asked to report any side effect experienced in the course of the study.
The maximum plasma concentration (Cmax) of SHR0302 | At protocol-specified times up to 72 hrs postdose
  Blood samples are taken on various timepoints to assess the pharmacokinetic parameters
The area under the plasma concentration-time curve (AUC) of SHR0302 | At protocol-specified times up to 72 hrs postdose
t1/2 of SHR0302 | At protocol-specified times up to 72 hrs postdose
Pharmacodynamics (PD)parameters of percent and actual change from baseline for a panel of JAK-dependent biomarkers | At protocol-specified times up to 24 hrs postdose
  To characterize the effects of SHR0302 on mechanism of action-related biomarkers in the blood over time - pharmacodynamics (PD) - in healthy volunteers.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Fourth Military Medical University, Xi’an, Shanxi, China